CLINICAL TRIAL: NCT05166616
Title: A Phase 1b Open-Label, Dose-Escalation, Safety, and Pharmacodynamic Study of Minnelide™ Capsules Given in Combination With Osimertinib in Patients With EGFR Mutated NSCLC
Brief Title: Minnelide and Osimertinib for the Treatment of Advanced EGFR Mutated Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20609; NCI-2021-12558 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20609 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2021-11-29; First posted 2021-12-22 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Advanced Lung Non-Small Cell Carcinoma; Locally Advanced Lung Non-Small Cell Carcinoma; Stage III Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8; Unresectable Lung Non-Small Cell Carcinoma
MeSH Terms: conditions — Lung Neoplasms | interventions — Biopsy; osimertinib; triptolide; 14-O-phosphonooxymethyltriptolide disodium salt

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (minnelide, osimertinib) (Experimental): Patients receive minnelide PO QD on days 1-21 and osimertinib PO QD on days 1-28. Cycles repeat every 28 days for 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Biopsy; Drug: Osimertinib; Drug: Triptolide Analog

INTERVENTIONS:
Procedure: Biopsy — Correlative studies
  Other Names: BIOPSY_TYPE; Bx
Drug: Osimertinib — Given PO
  Other Names: AZD-9291; AZD9291; Mereletinib; Tagrisso
Drug: Triptolide Analog — Given PO
  Other Names: Minnelide

SUMMARY:
This phase Ib trial tests the side effects and best dose of minnelide when given together with osimertinib for the treatment of non-small cell lung cancer that has spread to other places in the body (advanced) and has a change (mutation) in a gene called EGFR. Minnelide is a biologically inactive compound that can be broken down in the body to produce a drug that rapidly releases the active compound triptolide when exposed to phosphatases in the bloodstream. Sometimes, mutations in the EGFR gene cause EGFR proteins to be made in higher than normal amounts on some types of cancer cells. This causes cancer cells to divide more rapidly. Osimertinib may stop the growth of tumor cells by blocking EGFR that is needed for cell growth in this type of cancer. Minnelide and osimertinib may work better in treating patients with EGFR mutant advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) and the dose limiting toxicities (DLT) of triptolide analog (minnelide) capsules when given in combination with osimertinib.

II. To establish the dose of minnelide capsules recommended for future phase II studies when given in combination with full dose osimertinib (recommended phase II dose [RP2D]).

SECONDARY OBJECTIVES:

I. To observe patients for any evidence of antitumor activity of minnelide capsules by objective radiographic assessment when in combination with osimertinib.

II. To determine pharmacodynamic effects of minnelide capsules on heat shock protein (HSP)72 levels when given in combination with osimertinib.

EXPLORATORY OBJECTIVES:

I. Measure HSP levels, pre/post and during therapy as predictive biomarker. II. Determine levels of minnelide in the blood, and its effect. III. Determine the cell free deoxyribonucleic acid (DNA) in blood as biomarker. IV. Evaluate the microbiome pre-, during-, and post-therapy as potentiator of therapeutic response.

V. Determine the exosomes as biomarker.

OUTLINE: This is a dose-escalation study of minnelide.

Patients receive minnelide orally (PO) once daily (QD) on days 1-21 and osimertinib PO QD on days 1-28. Cycles repeat every 28 days for 6 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Agreement to two research biopsies

  * If tumor is unbiopsiable or not safely biopsied, exceptions may be granted with study principal investigator (PI) approval
* Age: >= 18 years
* Karnofsky performance >= 70%
* Histologically confirmed advanced non-small cell lung cancer (NSCLC). Patients with locally advanced NSCLC must not be candidates for surgical resection, radiation, or chemoradiation with curative intent
* The tumor harbors 1 of the 2 common epidermal growth factor receptor (EGFR) mutations known to be associated with epidermal growth factor receptor tyrosine kinase inhibitors (EGFR-TKI) sensitivity (Ex19del or L858R), either alone or in combination with other epidermal growth factor receptor (EGFR) mutations, which may include T790M
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Tumor progression after receiving standard/approved osimertinib
* Fully recovered from the acute toxic effects (except alopecia) to =< grade 1 to prior anti-cancer therapy. Grade 2 neuropathy is allowed
* Absolute neutrophil count (ANC) >= 1,500/mm^3 (within 14 days prior to day 1 of protocol therapy)

  * NOTE: Growth factor is not permitted within 14 days of ANC assessment
* Platelets >= 100,000/mm^3 (within 14 days prior to day 1 of protocol therapy)

  * NOTE: Platelet transfusions are not permitted within 14 days of platelet assessment
* Hemoglobin >= 9 g/dL (within 14 days prior to day 1 of protocol therapy)
* Total bilirubin =< 1.5 X ULN (unless has Gilbert's disease). Total bilirubin < 3 x ULN in the presence of documented Gilbert's disease (within 14 days prior to day 1 of protocol therapy)
* Aspartate aminotransferase (AST) =< 2.5 x upper limit of normal (ULN) (if liver metastases are present, then =< 5 x ULN is allowed) (within 14 days prior to day 1 of protocol therapy)
* Alanine aminotransferase (ALT) =< 2.5 x ULN if liver metastases are present, then =< 5 x ULN is allowed) (within 14 days prior to day 1 of protocol therapy)
* Alkaline phosphatase =< 2.5 x ULN if liver metastases are present, then =< 5 x ULN is allowed) (within 14 days prior to day 1 of protocol therapy)
* Serum creatinine within normal limits, OR creatinine clearance of >= 60 mL/min per 24 hour urine test for patients with creatinine levels above ULN (within 14 days prior to day 1 of protocol therapy)

  * Creatinine clearance (CrCl, by Cockcroft-Gault) is utilized for all patients to allow for evaluation of the effect of CrCl on the minnelide/triptolide exposures
* If not receiving anticoagulants: International normalized ratio (INR) OR prothrombin time (PT) =< 1.5 x ULN (within 14 days prior to day 1 of protocol therapy)

  * If on anticoagulant therapy: PT must be within therapeutic range of intended use of anticoagulants
* If not receiving anticoagulants: Activated partial thromboplastin time (aPTT) =< 1.5 x ULN (within 14 days prior to day 1 of protocol therapy)

  * If on anticoagulant therapy: aPTT must be within therapeutic range of intended use of anticoagulants
* Albumin >= 3.0 /dL (within 14 days prior to day 1 of protocol therapy)
* Urinalysis - no clinically significant abnormalities (within 14 days prior to day 1 of protocol therapy)
* QT corrected (QTc) =< 470 ms (using the Bazett's formula)

  * Note: To be performed within 28 days prior to Day 1 of protocol therapy.
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test (within 14 days prior to day 1 of protocol therapy)

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 6 weeks after the last dose of protocol therapy. Contraception must be continued following discontinuation of the study drugs for at least five half-lives of both study drugs

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)
  * Female patients of childbearing potential must:

    * Agree to practice 1 highly effective method of non-hormonal contraception and one additional effective (barrier) method at the same time, from the time of signing the informed consent through 180 days after the last dose of study drug, or
    * Agree to practice true abstinence, when is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g. calendar, ovulation, symptothermal, postovulation methods], withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together.)
    * Agree not to donate eggs (ova) during the course of this study or 180 days after receiving their last dose of study drug. Agree not to breast-feed for the duration of treatment through 6 months post treatment.
  * Male patients of childbearing potential must:

    * Agree to practice effective barrier contraception during the entire study treatment period and through 180 days after the last dose of study drug, or
    * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g. calendar, ovulation, symptothermal, postovulation methods for the female partner] and withdrawal are not acceptable methods of contraception. Female and male condoms should not be used together.)
    * Agree not to donate sperm during the course of this study or within 180 days after receiving their last dose of study drug.
* Patients must be able to swallow and retain oral medications
* Previously tolerant of osimertinib at 80 mg QD

Exclusion Criteria:

* Treatment with radiation therapy, surgery, chemotherapy, or investigational therapy within 21 days prior to day 1 of protocol therapy (6 weeks for nitrosoureas or Mitomycin C). Exceptions to this exclusion are brain radiation and osimertinib
* Biological therapy, immunotherapy within 21 days prior to day 1 of protocol therapy
* Strong CYP3A4 inducers/ inhibitors within 14 days prior to day 1 of protocol therapy
* Patients receiving class 1A or class III antiarrhythmic agents within 14 days prior to Day 1 of protocol therapy
* Herbal and alternative (eg. turmeric, cannabidiol, ginseng) medications within 7 days prior to Day 1 of protocol therapy
* Clarithromycin, loperamide, ondansetron within 7 days prior to day 1 of protocol therapy
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent
* Active diarrhea
* Clinically significant uncontrolled illness
* Known history of immunodeficiency virus (HIV) or hepatitis B or hepatitis C infection
* Prior malignancy other than carcinoma in situ of the cervix, or nonmelanoma skin cancer, unless that prior malignancy was diagnosed and definitively treated 5 or more years prior to study entry with no subsequent evidence of recurrence. Patients with a history of low grade (Gleason score =< 6 = Gleason Group 1) localized prostate cancer will be eligible even if diagnosed less than 5 years prior to study entry
* Females only: Pregnant or breastfeeding
* Any malabsorption condition
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures.
* New York Heart Association Class III or IV, cardiac disease, myocardial infarction within the past 6 months, unstable arrhythmia, or evidence of ischemia on electrocardiogram (ECG)
* Clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have previously-treated CNS metastases, are asymptomatic, and have had no requirement for steroid medication for 1 week prior to the first dose of study drug and have completed radiation 2 weeks prior to the first dose of study drug
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
* Diagnosis of congenital long QT syndrome
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2027-10-28 (Estimated); Study Completion 2027-10-28 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of osimertinib and minnelide | Up to 28 days
Recommended phase II dose (RP2D) of minnelide and osimertinib | Up to 28 days

SECONDARY OUTCOMES:
Pharmacodynamic effects of minnelide on heat shock protein (HSP)72 expression | Up to 2 years
  To analyze the pharmacodynamic effects of Minnelide on HSP72 protein levels in serum collected at specific timepoints before and after treatment.
Objective response rate | Up to 2 years
  Assessed per Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1.
Duration of overall response | Up to 2 years
Evidence of anti-tumor activity of minnelide when in combination with osimertinib | Up to 2 years
  Assessed by objective radiographic assessment.
Incidence of adverse events | Up to 2 years
  Assessed per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Progression-free survival (PFS) | Up to 2 years
  Assessed per RECIST v 1.1. Median PFS will be determined using the Kaplan-Meier method.
Overall survival | From the date of study enrollment to the date of death from any cause, assessed up to 2 years
  Assessed per RECIST v 1.1.

OTHER OUTCOMES:
HSP levels pre and post therapy | Baseline and up to 2 years
Levels of minnelide in the blood | Up to 2 years
Cell free deoxyribonucleic acid (DNA) in blood | Up to 2 years
Evaluation of the microbiome | Up to 2 years
  To evaluate the microbiome through amplicon sequencing of DNA extracted from fecal material collected by patients at baseline, restaging (2 cycles/8 weeks), and post-therapy (after disease progression/treatment discontinuation).
Determination of the exosomes | Up to 2 years
  To determine potential biomarkers through whole exome sequencing of tumor specimen. In brief, whole exome sequencing using a structured exome design will be performed on paired tumor/normal samples.
  This assay enables identification of mutations within exons as well as detection of structural variants including copy number variants and translocation breakpoints.

CONTACTS AND LOCATIONS:
Overall Officials: Erminia Massarelli, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States